CLINICAL TRIAL: NCT03599609
Title: Central Nervous System Vascular Changes Evidenced by Magnetic Resonance Imaging in Adult Patients With Sickle Cell Disease and the Effect of Treatment With Simvastatin
Brief Title: Central Nervous System Vascular Changes in Adult Sickle Cell Disease and the Effect of Treatment With Simvastatin
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Bruno Deltreggia Benites, Principal Investigator, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2.487.922
Record Dates: First submitted 2018-07-02; First posted 2018-07-26 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Sickle Cell Disease; Stroke
MeSH Terms: conditions — Anemia, Sickle Cell; Stroke | interventions — Simvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Treatment: Simvastatin 40mg/day
  Interventions: Drug: Simvastatin 40mg

INTERVENTIONS:
Drug: Simvastatin 40mg — Simvastatin 40mg, once daily

SUMMARY:
Stroke is a frequent complication of sickle cell disease (SCD), with varying levels of central nervous system (CNS) involvement. The summation of several ischemic events, even when silent, can lead to devastating consequences, from reduced academic performance to physical dependence. Despite knowledge that brain flow velocities evaluated by Doppler ultrasound identify pediatric SCD patients at a greater stroke risk (Adams et al, NEJM 1998; 339:5-11), this method is not able to predict the occurrence of strokes in adults. There is also no consensus on the management of adult patients in relation to primary and secondary prevention. The aim of this study is to evaluate the effects of the administration of Simvastatin on CNS structural and functional vascular changes in 30 adult patients with SCD (SS and Sβ), above 35 years of age, observed through Magnetic Resonance Imaging (MRI). The data on the effect of simvastatin on disease manifestations is quite scarce, however this drug reportedly significantly reduces plasma concentrations of adhesion molecules and inflammatory markers, such as E-selectin, VEGF, CRP and IL-6 (Hoppe et al, BJH 2011; 153:655-663; Hoppe et al, BJH 2017;177:620-629). Thus, in addition to the search for early diagnostic markers and risk stratification for primary or recurrent stroke, we will also compare CNS images before and 12 months after the administration of Simvastatin. The drug alter stroke recurrence rates in the general adult population, but their effects on vascular changes in patients with SCD have not yet been adequately elucidated. This is particularly important because these are low cost drugs which present good tolerability, and could be part of the therapeutic arsenal of SCD, even in low income settings. Concomitantly with the CNS evaluation, this study also intends to investigate molecular pathways that may be affected by the drugs. We will evaluate microvesicle release patterns, as well as the content of microRNAs possibly involved in the occurrence of stroke, in addition to metabolomic studies and plasma cytokine profile.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Sickle Cell Disease

Exclusion Criteria:

* Previous stroke
* Some relevant concomitant clinical condition (cancer, AIDS, inflammatory / autoimmune diseases, etc.).
* Pregnancy
* Individuals considered to be vulnerable (minors,institutionalized individuals, patients with a history of psychiatric illness with cognitive impairment or incapacity)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Stroke prevention | 5 years
  Number of patients in the cohort presenting srtoke or silent infarction detected at MRI

SECONDARY OUTCOMES:
Improvement of hemodynamic parameters in MRI:velocity | 1 year
  Evaluation of changes in vessel segment-averaged velocity (cm/s) in the Circle of Willis
Improvement of hemodynamic parameters in MRI: lumen area | 1 year
  Evaluation of changes in vessel lumen area (mm2) in the Circle of Willis
Improvement of hemodynamic parameters in MRI: flow | 1 year
  Evaluation of changes in flow (ml/s) in the Circle of Willis
Improvement of hemodynamic parameters in MRI: endothelial shear stress | 1 year
  Evaluation of changes in endothelial shear stress (Pa) in the Circle of Willis

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Benites, MD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Hematology and Transfusion Medicine Center, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No